CLINICAL TRIAL: NCT05294757
Title: Development of Continuous Assessment of Muscle Quality and Frailty in Older Subjects Using Multi-parametric Combinations of Ultrasound and Blood Biomarkers: a Study Protocol for a Quasi-experimental Multi-center Study (ECOFRAIL Study)
Brief Title: Development of Continuous Assessment of Frailty and Muscle Quality in Older Subjects: ECOFRAIL Protocol
Acronym: ECOFRAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Deusto (Other)
Collaborators: Complejo Hospitalario Universitario de Albacete (Other); Biogipuzkoa Health Research Institute (Other); Hospital Universitario Getafe (Other); European University of Vitoria-Gasteiz (Other)
Responsible Party: Principal Investigator, Xabier Rio de Frutos, Researcher HealthPASS team, University of Deusto
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECOFRAIL
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Frailty; Sarcopenia; Ultrasonography; Exercise
Keywords: Echography; Biomarkers; Diagnostic; Muscle; Exercise
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity; Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: three groups: control, exercise, and fragile
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hospital control (No Intervention): Hospital control cohort: Participants will be consecutively recruited from the scheduled patient list of the frailty unit, day hospital, and the outpatient clinic of the Geriatrics Department of Hospital 2. After obtaining informed consent, baseline study variables will be collected. Patients will be followed-up for a 16-week period, under usual care. After the follow-up period, baseline evaluation will be repeated.
- Exercise (Experimental): Elderly people without muscle problems participating in the exercise program to see improvements in their muscle mass levels and quality
  Interventions: Other: Physical exercise
- Primary care Control (No Intervention): Primary care cohort: Participants will be consecutively recruited from the scheduled patient list of the Primary Care Units. After informed consent acquisition, baseline study variables will be collected. Patients will be followed-up during one year, under usual care. After the one-year follow-up, the baseline evaluation will be repeated.

INTERVENTIONS:
Other: Physical exercise — 1. Hospital exercise cohort: Participants will be consecutively recruited from the scheduled patient list of the falls unit and the outpatient clinics of Hospital 1. After informed consent acquisition, patients will receive a baseline clinical evaluation. Ultrasound measurements and DXA scan will be conducted, and blood samples will be collected, processed, and stored. Patients will be included in the 16-week multicomponent physical exercise program described below. After the completion of the exercise program, at 16-week follow-up, clinical evaluation, ultrasound, DXA, and blood-sample testing will be repeated.
  Arms: Exercise

SUMMARY:
We are conducting a study in different centers in Spain in elderly people, in order to assess the effectiveness of a physical exercise intervention program in people in a situation of frailty. Frailty in an elderly person is a situation in which, although there are no major differences in their usual abilities, the person presents a certain decrease in their capacities. This slight decrease is usually accompanied by a progressive deterioration.

DETAILED DESCRIPTION:
Background: Frailty derived from muscle quality loss can potentially be delayed through early detection and physical exercise interventions. There is a need for affordable tools for the objective evaluation of muscle quality, in both cross-sectional and longitudinal assessment. Literature suggests that quantitative analysis of ultrasound data captures morphometric, compositional and microstructural muscle properties, while biological essays derived from blood samples are associated with functional information. The aim of this study is to evaluate multi-parametric combinations of ultrasound and blood-based biomarkers to provide a cross-sectional evaluation of the patient frailty phenotype and to monitor muscle quality changes associated with supervised exercise programs.

Methods: This is a prospective observational multi-center study including patients older than 70 years with ability to give informed consent. We will recruit 100 patients from hospital environments and 100 from primary care facilities. At least two exams per patient (baseline and follow-up), with a total of (with a minimum total of 400 exams) exams. In the hospital environments, 50 patients will be measured pre/post a 16-week individualized and supervised exercise programme, and 50 patients will be followed-up after the same period without intervention. The primary care patients will undergo a one-year follow-up evaluation. The primary goal is to compare cross-sectional evaluations of physical performance, functional capacity, body composition and derived scales of sarcopenia and frailty with biomarker combinations obtained from muscle ultrasound and blood-based essays. We will analyze ultrasound raw data obtained with a point-of-care device, and a set of biomarkers previously associated with frailty by quantitative Real time PCR (qRT-PCR) and enzyme-linked immunosorbent assay (ELISA). Secondly, we will analyze the sensitivity of these biomarkers to detect short-term muscle quality changes as well as functional improvement after a supervised exercise intervention with respect to usual care.

Discussion: The presented study protocol will combine portable technologies based on quantitative muscle ultrasound and blood biomarkers for objective cross-sectional assessment of muscle quality in both hospital and primary care settings. It aims to provide data to investigate associations between biomarker combinations with cross-sectional clinical assessment of frailty and sarcopenia, as well as musculoskeletal changes after multicomponent physical exercise programs.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 70 years old.
2. Either gender.
3. Ability to provide informed consent.
4. Ability to perform all the functional tests.
5. In the hospital exercise cohort, ability to perform the physical exercise program.

Exclusion Criteria:

1. Expected survival inferior to one year.
2. Barthel scale < 70.
3. Moderate to severe cognitive impairment.
4. Refuse to participate.
5. Medical conditions that may condition or difficult the follow-up assessments.
6. Older adults already included in regular physical exercise programmes will be excluded to participate in the hospital exercise cohort.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker - Quality of Life - Muscle mass | 2 years
  Association between quantitative ultrasound biomarkers associated to muscle mass and quality and extracted from raw data and blood-based biomarkers and combinations thereof with clinical variables including frailty, sarcopenia, physical function, disability, nutritional status, body composition, and Quality of Life in three cohorts of older adults: hospital control cohort, hospital exercise cohort, and primary care cohort.
  Muscle quality and mass: Ultrasound. Thickness (mm), cross-sectional area (cm²), perimeter (mm) and pennation angle (°). Frailty: FRAIL scale range 0-5. Frailty phenotype (0-5). Sarcopenia: SARC-F scale (0-10). Disability: GDS, 7 stages. Barthel index (0-100). Lawton and Brody index 0-8. Physical function: SPPB (0-12). IPAQ (0-3). Gait speed test, seconds. Grip strength, Jamar dynamometer, kilograms.
  Quality of life: EQ 5D-5L, scale of 0-100.
  Blood biomarkers: Vitamin D, Lutein zeaxanthin, Troponin T, Pro-BNP, and sRAGE with ELISA, miRNAs (qRT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Sanabria, Ph.D., Principal Investigator — University of Deusto
Locations (3):
- Spain (3):
  - Complejo Hospitalario Universitario de Albacete, Albacete, Castille-La Mancha
  - Donostialdea, Osakidetza, Donostia / San Sebastian
  - Hospital Universitario de Getafe, Getafe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Virto N, Rio X, Angulo-Garay G, Garcia Molina R, Avendano Cespedes A, Cortes Zamora EB, Gomez Jimenez E, Alcantud Corcoles R, Rodriguez Manas L, Costa-Grille A, Matheu A, Marcos-Perez D, Lazcano U, Vergara I, Arjona L, Saeteros M, Lopez-de-Ipina D, Coca A, Abizanda Soler P, Sanabria SJ. Development of Continuous Assessment of Muscle Quality and Frailty in Older Patients Using Multiparametric Combinations of Ultrasound and Blood Biomarkers: Protocol for the ECOFRAIL Study. JMIR Res Protoc. 2024 Feb 23;13:e50325. doi: 10.2196/50325. PMID 38393761